CLINICAL TRIAL: NCT00556686
Title: Salivary Catecholamines in Aphthous Stomatitis
Brief Title: Salivary Catecholamines in Aphthous Stomatitis (Canker Sores)
Status: Withdrawn | Type: Observational
Why Stopped: We are currently modifying the study
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200614581
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Canker Sore
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Individuals with a history of canker sores.
- 2: Individuals with no history of canker sores.

SUMMARY:
The purpose of this study is to examine how compounds produced in patients with canker sores affect wound healing.

DETAILED DESCRIPTION:
The purpose of this study is to determine if salivary catecholamines are elevated in patients with the disease aphthous stomatitis. The results of this study will be combined with those performed in collaboration with a co-Investigator to understand the effects of catecholamines on mucosal wound healing and oral epithelial cell migration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older, both genders
* History of recurrent aphthous ulcers with 4 or more episodes per year

Exclusion Criteria:

* History of salivary gland disease including Sjogren's disease, parotitis, and sialolithiasis
* History of benign or malignant salivary gland tumor
* History of celiac disease, ulcerative colitis or Crohn's disease
* Patients on medications that affect salivary flow such as anti-depressants and anti-cholinergic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will be sampled from the community.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Fazel, MD, DDS, Principal Investigator — University of California, Davis

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical